CLINICAL TRIAL: NCT06284473
Title: Intranasal Ketamine as a Supplement to Local Anesthesia to Reduce Pain Associated With Minor Procedures in the Emergency Department
Brief Title: Ketamine as a Supplement to Local Anesthesia for Minor Procedures
Acronym: INK-MP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Trent Reed, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 212154
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pain, Procedural; Minor Laceration; Abscess
Keywords: IN Ketamine; Sub-dissociative dose; Minor procedure
MeSH Terms: conditions — Pain, Procedural; Abscess | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients presenting to the emergency department at Loyola University Medical Center for a minor medical procedure requiring local anesthesia will be randomly assigned to receive either standard local anesthesia with 0.7 mg/kg intranasal ketamine before the procedure or to standard local anesthesia with volume-based dose saline before the procedure using a 1:1 random block allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and study personnel are blinded except for the clinical pharmacist who prepares the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Ketamine (Experimental): Participants assigned to this arm will receive intranasal ketamine administered at 0.7mg/kg along with normal lidocaine local sedation
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Participants assigned to this arm will receive volume-based dose of intranasal saline administered along with normal lidocaine local sedation
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ketamine — Ketamine is an N-methyl-D aspartate receptor agonist
  Arms: Intranasal Ketamine
Other: Saline — Intranasal saline flushes pollen, dust, and other debris from nasal passages. It also removes excess mucus and adds moisture
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This trial is a double-blind randomized controlled clinical trial of adults and children (ages 7 to less than 70 years). Patients who present to the ED and who undergo minor bedside procedures that require local anesthesia will be divided into two groups: The first group will be treated with 0.7 mg/kg intranasal ketamine as well as standard local anesthesia for the procedure (treatment cohort). The second group will be treated with a volume-based dose of intranasal saline solution as well as standard local anesthesia for the procedure (control cohort). The primary aim is to assess whether patients in the treatment cohort report lower pain scores on the Numerical Rating Scale (NRS-100) when compared to patients in the control cohort. For adult patients, a secondary aim is to compare agitation between the two cohorts using the Richmond Agitation Sedation Scale (RASS) and, for pediatric patients, a secondary aim is to compare alertness between the two cohorts using the University of Michigan Sedation Scale (UMSS).

Results obtained from specific procedures will be analyzed on a spectrum of complexity and general length of recovery time. Scientific achievements may include finding a safe and effective way to reduce pain and discomfort during minor procedures in the Emergency Department. Additionally, it would provide opportunities for more research on sub-dissociative doses of ketamine during minor procedures: a topic in which there is still a gap in the published research

DETAILED DESCRIPTION:
Patient experiences in the emergency department (ED) are commonly painful and uncomfortable, particularly when patients must undergo procedures. Managing acute pain and procedural pain for minor procedures in the ED can be challenging. Ketamine is an N-methyl-D aspartate receptor agonist gaining popularity in clinical settings and has also been shown in several studies to potentially treat depression. Several randomized clinical studies have shown that ketamine is a comparable pain relief medication to opioid analgesics in both acute pain and traumatic settings. Its uses for pain control in the ED have been extensively studied with evidence supporting its safety and efficacy. Ketamine can be administered in different ways including intravenously and intranasally. Intravenously, doses above 1 mg/kg of ketamine can induce dissociation- this dose is commonly used for procedural sedation. At lower doses, specifically sub-dissociative doses, ketamine (SDK) acts to alleviate pain (cancerous, neuropathic, and perioperative). Trials using intravenous SDK suggest efficacy similar to traditional intravenous opioid analgesics.

SDK is currently being utilized by emergency medicine physicians in the ED for pain control in doses up to 0.3 mg/kg intravenously and up to 1 mg/kg intranasally. Additionally, the use of SDK in the ED is also supported by the American College of Emergency Physicians. While the literature has extensively documented and supported the safety and efficacy of SDK, there is a gap in the literature for its use in the management of pain for minor procedures in the ED. Intranasal ketamine may be a valuable supplement to standard medical treatment in procedures that would not normally require intravenous access. Minor procedures requiring local anesthesia performed in the ED can still be painful including but not limited to suturing, incision and drainage of an abscess, and digital blocks. Traditionally, many of these procedures are completed using only local anesthesia. Soft tissue and/or very large abscess are sometimes not alleviated by local anesthesia alone. The use of intranasal ketamine to alleviate pain during these and other painful procedures may provide patients with more comfort and pain relief than local anesthesia alone. Dosing for chronic pain and acute pain differ in that chronic pain typically requires higher doses than acute pain. Side effects are related to ketamine dosage and administration type. Thus, patients treated for chronic pain with higher doses of SDK often experience more side effects than patients with acute pain treated with lower doses of SDK. Additionally, compared to placebo and opioid groups in various studies, ketamine was associated with greater risk of neurological, psychological, and minor cardiologic effects. However, the opioid groups typically had a higher risk for major cardiopulmonary effects. The most common side effect of intranasal SDK are bad taste in the mouth, dizziness, and sleepiness. A dose of 0.7 mg/kg IN ketamine has been determined to be a suitable analgesic dose for patients with pain in the ED. While studies have shown the efficacy and safety of using ketamine for pain control, no studies to date have looked at its possible use to decrease pain during minor procedures in the ED.

The investigators aim to determine if a sub-dissociative dose of 0.7 mg/kg intranasal ketamine is a desirable choice to reduce pain associated with minor procedures requiring local anesthesia in the ED. These procedures include incision and drainage of an abscess, laceration repairs requiring sutures, nerve blocks (specifically digital nerve blocks), and other minor procedures requiring local anesthesia. The investigators hypothesize that adult and pediatric patients presenting to the ED and undergoing painful minor procedures will report lower pain scores when treated with 0.7 mg/kg intranasal ketamine in addition to standard local anesthesia than patients who receive a volume-based dose of saline solution with standard local anesthesia (control). Additionally, the investigators hypothesize that patients in the treatment cohort will report few side-effects as measured by the Richmond Agitation Sedation Scale (RASS)(i.e., for adult patients) or University of Michigan Sedation Scale (UMSS) (i.e., for pediatric patients). The minor procedures listed above typically require the use of local anesthesia but do not typically require intravenous access. Thus, the use of intranasal ketamine instead of intravenous analgesia minimizes the changes that would be made to the current standard of carrying out these procedures.

In order to avoid a potential confounder of variation in baseline pain severity of the different procedures, only patients undergoing minor procedures that have a similar pain profile will be randomized. Additional aims of the study include decreasing perceived agitation using RASS or UMSS. Collecting data on pain and total discomfort using the NRS-100 point pain scale will provide a unidimensional measurement of patients' subjective interpretation of their pain. The investigators hope to demonstrate that using ketamine at 0.7 mg/kg for associated pain during minor procedures is efficacious and minimizes adverse side effects of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Minor Procedure in the ED
* Weight not to exceed 115kg

Exclusion Criteria:

* Altered Mental Status
* Pregnancy
* Breastfeeding
* Acute head or eye injury
* Intercranial Hypertension
* Hx of seizures
* Hx of chronic pain
* Unstable vital signs
* Allergy to Ketamine
* Hepatic or Renal Insufficiency
* Hx of Psychiatric Illness
* Hx of alcohol/drug abuse

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Immediate pain | 15 minutes
  Pain will be measured using the numeric rating scale which is a scale ranging from 0 to 100, where higher values report greater pain
Acute pain | 30 minutes
  Pain will be measured using the numeric rating scale which is a scale ranging from 0 to 100, where higher values report greater pain
Delayed pain | 60 minutes
  Pain will be measured using the numeric rating scale which is a scale ranging from 0 to 100, where higher values report greater pain

SECONDARY OUTCOMES:
Immediate agitation | 15 minutes
  For adults, agitation will be measured using the Richmond Agitation Sedation Scale (RASS) which is a 10-point scale (range: -5 to +4), where higher scores reflect greater agitation.
Acute agitation | 30 minutes
  For adults, agitation will be measured using the Richmond Agitation Sedation Scale (RASS) which is a 10-point scale (range: -5 to +4), where higher scores reflect greater agitation.
Delayed agitation | 60 minutes
  For adults, agitation will be measured using the Richmond Agitation Sedation Scale (RASS) which is a 10-point scale (range: -5 to +4), where higher scores reflect greater agitation.
Immediate alertness | 15 minutes
  For pediatric patients, agitation will be measured using the University of Michigan Sedation Scale (UMSS) which assesses the level of alertness on a five-point scale ranging from 0 (awake and alert) to 4 (unarousable).
Acute alertness | 30 minutes
  For pediatric patients, agitation will be measured using the University of Michigan Sedation Scale (UMSS) which assesses the level of alertness on a five-point scale ranging from 0 (awake and alert) to 4 (unarousable).
Delayed alertness | 60 minutes
  For pediatric patients, agitation will be measured using the University of Michigan Sedation Scale (UMSS) which assesses the level of alertness on a five-point scale ranging from 0 (awake and alert) to 4 (unarousable).

CONTACTS AND LOCATIONS:
Overall Officials: Trent Reed, DO, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers

REFERENCES:
- [Background] Shimonovich S, Gigi R, Shapira A, Sarig-Meth T, Nadav D, Rozenek M, West D, Halpern P. Intranasal ketamine for acute traumatic pain in the Emergency Department: a prospective, randomized clinical trial of efficacy and safety. BMC Emerg Med. 2016 Nov 9;16(1):43. doi: 10.1186/s12873-016-0107-0. PMID 27829367
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Background] Zekry O, Gibson SB, Aggarwal A. Subanesthetic, Subcutaneous Ketamine Infusion Therapy in the Treatment of Chronic Nonmalignant Pain. J Pain Palliat Care Pharmacother. 2016 Jun;30(2):91-8. doi: 10.3109/15360288.2016.1161690. Epub 2016 Apr 19. PMID 27092576
- [Background] Hanna AF, Armstrong JS, Smith AJ. Effects of Intravenous Ketamine Infusions in a Neuropathic Pain Patient with Lichen Sclerosus et Atrophicus. Case Rep Dermatol. 2016 Jun 6;8(2):164-70. doi: 10.1159/000446528. eCollection 2016 May-Aug. PMID 27462225
- [Background] Miller JP, Schauer SG, Ganem VJ, Bebarta VS. Low-dose ketamine vs morphine for acute pain in the ED: a randomized controlled trial. Am J Emerg Med. 2015 Mar;33(3):402-8. doi: 10.1016/j.ajem.2014.12.058. Epub 2015 Jan 7. PMID 25624076
- [Background] Karlow N, Schlaepfer CH, Stoll CRT, Doering M, Carpenter CR, Colditz GA, Motov S, Miller J, Schwarz ES. A Systematic Review and Meta-analysis of Ketamine as an Alternative to Opioids for Acute Pain in the Emergency Department. Acad Emerg Med. 2018 Oct;25(10):1086-1097. doi: 10.1111/acem.13502. Epub 2018 Jul 17. PMID 30019434
- [Background] Optimizing the Treatment of Acute Pain in the Emergency Department. Ann Emerg Med. 2017 Sep;70(3):446-448. doi: 10.1016/j.annemergmed.2017.06.043. No abstract available. PMID 28844277
- [Background] Payne CG, Edbrooke DL, Davies GK. Minor procedures in the accident and emergency department: can Entonox help? Arch Emerg Med. 1991 Mar;8(1):24-32. doi: 10.1136/emj.8.1.24. PMID 1854389
- [Background] Allen CA, Ivester JR Jr. Ketamine for Pain Management-Side Effects & Potential Adverse Events. Pain Manag Nurs. 2017 Dec;18(6):372-377. doi: 10.1016/j.pmn.2017.05.006. Epub 2017 Jul 23. PMID 28743507
- [Background] Lee EN, Lee JH. The Effects of Low-Dose Ketamine on Acute Pain in an Emergency Setting: A Systematic Review and Meta-Analysis. PLoS One. 2016 Oct 27;11(10):e0165461. doi: 10.1371/journal.pone.0165461. eCollection 2016. PMID 27788221
- [Background] Reynolds SL, Studnek JR, Bryant K, VanderHave K, Grossman E, Moore CG, Young J, Hogg M, Runyon MS. Study protocol of a randomised controlled trial of intranasal ketamine compared with intranasal fentanyl for analgesia in children with suspected, isolated extremity fractures in the paediatric emergency department. BMJ Open. 2016 Sep 8;6(9):e012190. doi: 10.1136/bmjopen-2016-012190. PMID 27609854
- [Background] Shrestha R, Pant S, Shrestha A, Batajoo KH, Thapa R, Vaidya S. Intranasal ketamine for the treatment of patients with acute pain in the emergency department. World J Emerg Med. 2016;7(1):19-24. doi: 10.5847/wjem.j.1920-8642.2016.01.003. PMID 27006733
- [Background] Reynolds SL, Bryant KK, Studnek JR, Hogg M, Dunn C, Templin MA, Moore CG, Young JR, Walker KR, Runyon MS. Randomized Controlled Feasibility Trial of Intranasal Ketamine Compared to Intranasal Fentanyl for Analgesia in Children with Suspected Extremity Fractures. Acad Emerg Med. 2017 Dec;24(12):1430-1440. doi: 10.1111/acem.13313. Epub 2017 Nov 3. PMID 28926159
- [Background] Bouida W, Bel Haj Ali K, Ben Soltane H, Msolli MA, Boubaker H, Sekma A, Beltaief K, Grissa MH, Methamem M, Boukef R, Belguith A, Nouira S. Effect on Opioids Requirement of Early Administration of Intranasal Ketamine for Acute Traumatic Pain. Clin J Pain. 2020 Jun;36(6):458-462. doi: 10.1097/AJP.0000000000000821. PMID 32080000